CLINICAL TRIAL: NCT01110902
Title: A 8-week, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multi-center Study of the Efficacy and Safety of Agomelatine 0.5 mg and 1 mg Sublingual Tablets Administered Once Daily in Patients With Major Depressive Disorder (MDD)
Brief Title: Efficacy, Safety and Tolerability of Agomelatine Sublingual Tablets in the Treatment of Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAGO178C2302
Record Dates: First submitted 2010-04-23; First posted 2010-04-27 (Estimated); Last update posted 2020-12-24 (Actual); Status verified 2012-09

CONDITIONS: Major Depressive Disorder
Keywords: Agomelatine; Major Depressive Disorder; MDD; depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — agomelatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- AGO178C 0.5 mg /day (Experimental)
  Interventions: Drug: Agomelatine (AGO178C)
- AGO178C 1 mg / day (Experimental)
  Interventions: Drug: Agomelatine (AGO178C)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Agomelatine (AGO178C)
  Arms: AGO178C 0.5 mg /day; AGO178C 1 mg / day
Drug: Placebo
  Arms: Placebo

SUMMARY:
The study will assess efficacy, safety and tolerability of 0.5 mg/day and 1 mg/day of sublingual (under the tongue) formulation of agomelatine in patients with Major Depressive Disorder. This study includes an 8-week double-blind phase.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of MDD, single or recurrent episode, according to DSM-IV criteria.
* Current episode ≥4 weeks.
* CGI-Severity score ≥4 at Screening and Baseline.

Exclusion Criteria:

* History of bipolar disorder (I or II), schizophrenia, schizoaffective disorder, eating disorder (current or during previous one year), obsessive-compulsive disorder.
* Any other current Axis I disorder other than MDD which is the focus of treatment.
* Substance or alcohol abuse in the last 30 days, dependence in the last 6 months.
* Concomitant psychotropic medication, including herbal preparations and melatonin.
* Psychotherapy of any type.
* Prior exposure to agomelatine.
* Female patients of childbearing potential who are not using effective contraception.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 589 (Actual)
Dates: Start 2010-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to endpoint at Week 8 using the total score of the Hamilton Depression Rating Scale | Baseline and 8 weeks

SECONDARY OUTCOMES:
Effect on subjective sleep, as measured by the score of the Leeds Sleep Evaluation Questionnaire (LSEQ) domain "quality of sleep" at Week 8 | 8 weeks
Proportion of patients who demonstrate clinical response, where response is defined by a reduction of at least 50% in the Baseline clinician-rated HAM-D total score at Week 8 endpoint | 8 weeks
Proportion of patients who demonstrate clinical improvement at Week 8, where improvement is defined by a score of 1 or 2 on the CGI-I scale | 8 weeks
Proportion of patients who achieve remission | 8 weeks
Safety and tolerability by adverse events and serious adverse events, and assessment of suicidal ideation and behavior by Columbia Suicide Severity Rating Scale. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (45):
- United States (43):
  - University of Alabama at Birmingham, Department of Psychiatry, Birmingham, Alabama
  - ATP Clinical Research, Costa Mesa, California
  - Valley Clinical Research, El Centro, California
  - Collaborative Neuroscience Network, Garden Grove, California
  - University of California, Irvine Medical Center, Orange, California
  - Anderson Clinical Research, Redlands, California
  - Affiliated Research Institute, San Diego, California
  - California Neuroscience Research Medical Group, Inc., Sherman Oaks, California
  - Viking Clinical Research, Temecula, California
  - ICSL Clinical Studies, Altamonte Springs, Florida
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Arocha Research Center, Coral Gables, Florida
  - Innova Clinical Trials, Miami, Florida
  - Miami Research Associates, South Miami, Florida
  - Emory University, Atlanta, Georgia
  - Alexian Brothers Center for Psychiatric Research, Hoffman Estates, Illinois
  - Joliet Center for Clinical Research, Joliet, Illinois
  - CNS Clinical Trials, Park Ridge, Illinois
  - Deaconess Clinic, Evansville, Indiana
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Pharmasite Research, Pikesville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Clinical Trials, Brighton, Massachusetts
  - Mercy Health Research, St Louis, Missouri
  - Premier Psychiatry Group, LLC, Lincoln, Nebraska
  - CRI Worldwide, LLC - Lourdes Division, Willingboro, New Jersey
  - Social Psychiatric Research Institute, Brooklyn, New York
  - Eastside Comprehensive Medical Service, New York, New York
  - Neurobehavioral Clinical Research, Canton, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Neurology & Neuroscience Center of Ohio, Toledo, Ohio
  - SP Research, Oklahoma City, Oklahoma
  - Willamette Valley Clinical Studies, Eugene, Oregon
  - Summit Research Network, Portland, Oregon
  - CRI Worldwide, LLC - Kirkbride Division, Philadelphia, Pennsylvania
  - Medical University of South Carolina, North Charleston, South Carolina
  - CNS Healthcare, Memphis, Tennessee
  - Research Strategies, Memphis, Tennessee
  - FutureSearch Trials, Austin, Texas
  - Claghorn-Lesem Research Clinic, Inc., Houston, Texas
  - University of Utah, Department of Psychiatry, Salt Lake City, Utah
  - Northwest Clinical Research Center, Bellevue, Washington
  - Summit Research, Seattle, Washington
- Puerto Rico (2):
  - Caribbean Research and Education Center, Bayamón
  - Dharma Institute and Research Center, San Juan

REFERENCES:
- See also: Results for CAGO178C2302 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=6523
- See also: Click here for more information about this study: — http://novartisclinicaltrials.com